CLINICAL TRIAL: NCT00010465
Title: Osteopathic Manipulation and Echinacea for the Treatment of Recurrent Ear Infections in Children
Brief Title: Nervous System Manipulation and Botanicals for the Treatment of Recurrent Ear Infections in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: P50AT000008-01P1 (NIH); 1P50AT000008-01 (NIH); NCT00009269 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media

INTERVENTIONS:
Procedure: Craniosacral Osteopathic Manipulative Treatment
Drug: Botanicals

SUMMARY:
The purpose of this study is to determine the efficacy of echinacea therapy and osteopathic manipulation for the prevention of further ear infections in children with recurrent ear infections (otitis media).

DETAILED DESCRIPTION:
Acute otitis media (inflammation of the middle ear) occurs in 60% of infants during the first year of life and in 85% by age 3. Approximately 17% of children suffer recurrent otitis media during the first year of life. Following acute otitis media, middle ear fluid effusions can persist for weeks to months. Approximately 40% of children with middle ear effusions have mild to moderate hearing loss for the duration of the effusion, and several studies have found evidence for impaired speech and language development among children with prolonged middle ear effusion. Since antibiotic use has become widespread, concern has emerged regarding antibiotic resistant S. pneumoniae strains and other bacteria. Children with recurrent otitis media commonly receive prophylactic antibiotic therapy or surgical insertion of tubes to prevent accumulation of middle ear effusion. The prevalence of pediatric use of complementary alternative medical (CAM) approaches for prevention of otitis media has not been widely quantified. This study will evaluate the use of osteopathic manipulation and echinacea therapy to prevent ear infection in children with recurrent otitis media.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Aldous, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Derived] Wahl RA, Aldous MB, Worden KA, Grant KL. Echinacea purpurea and osteopathic manipulative treatment in children with recurrent otitis media: a randomized controlled trial. BMC Complement Altern Med. 2008 Oct 2;8:56. doi: 10.1186/1472-6882-8-56. PMID 18831749